CLINICAL TRIAL: NCT05843435
Title: Brain Connectivity Between Networks Implied in Inhibition and Cue-reactivity in Alcohol Use Disorder
Acronym: NIQA
Status: Completed | Type: Observational
Sponsor: University of Bern (Other)
Collaborators: Clinic Suedhang (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2023-00736
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Alcohol Use Disorder
Keywords: Inhibition, Psychology; Magnetic Resonance Imaging; Drinking Behavior
MeSH Terms: conditions — Alcoholism; Inhibition, Psychological; Drinking Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Alcohol Use Disorder/AUD: A group of 30 detoxified patients who are part of the specialized residential treatment program at the Clinic Suedhang in Kirchlindach in Switzerland.
  Interventions: Behavioral: Go-Nogo-task during functional magnetic resonance imaging; Other: Resting-state functional magnetic resonance imaging
- Healthy Controls/HC: A group of 30 age- and gender-matched healthy control subjects who are recruited via advertisement in social media or local newspaper.
  Interventions: Behavioral: Go-Nogo-task during functional magnetic resonance imaging; Other: Resting-state functional magnetic resonance imaging

INTERVENTIONS:
Behavioral: Go-Nogo-task during functional magnetic resonance imaging — Go-Nogo-task (GNG) implemented as a mixed block- and event-related design paradigm for task-related functional resonance imaging. It is composed of six blocks, each containing an event-related inhibitory control GNG. There are two blocks with an alcohol-related GNG, two blocks with a neutral GNG, and two blocks with a mixed GNG paradigm. The blocks are presented in a counterbalanced fashion between the participants. Each block contains 125 Go-trials and 25 NoGo-trials (ratio 5:1), resulting in 150 trials per block with a block time of 5 minutes. Participants are instructed to press a button whenever a stimulus appears on the screen (Go-trial). The only exception to this rule is when the same stimulus appears twice (NoGo-trial). Stimulus material consists of 60 alcohol-related and 60 neutral pictures, presented in a pseudo-randomized order.
  Other Names: Siemens Terra 7T
Other: Resting-state functional magnetic resonance imaging — An fMRI (multiband-echo-planar imaging) blood oxygenated level dependent (BOLD) protocol is run during 6 minutes of rest. This protocol allows the assessment of connectivity measures at rest, which can be compared to connectivity changes during the GNG task.

SUMMARY:
Research about patients with alcohol use disorder has shown that task-related brain activation patterns as well as resting-state connectivity (measured with functional magnetic resonance imaging) change with clinical parameters such as the extent of craving and duration of abstinence during treatment. These brain activation alterations are related to treatment success. Although an imbalance between increased cue-reactivity and impaired counteracting inhibitory control processes are at the core of most neuropsychological conceptualizations of alcohol use disorder, the direct interaction between these two processes has not yet been investigated. Therefore, the investigators aim to study patients with alcohol use disorder in an ultra-high-field 7 Tesla magnetic resonance imaging scanner to identify fine-grained activation and connectivity patterns. The investigators would like to improve the knowledge of the interplay between the brain networks for inhibition and cue-reactivity, as well as to explore its influence on craving and treatment success. The investigators hypothesize that a more pronounced negative relationship between increased cue-reactivity and reduced inhibitory control processes in the brain is linked to higher craving and worse relapse probability.

DETAILED DESCRIPTION:
Even if an imbalance between enhanced cue-reactivity and impaired opposing control processes is at the center of most neuroscientific conceptualizations of alcohol use disorder (AUD), these two processes are still rarely investigated in direct interaction.

Attempting to target both processes in one design, initial studies reported enhanced brain activation in anterior cingulate cortex (ACC) and ventrolateral prefrontal cortex (vlPFC), when control processes had to be carried out in the context of alcohol-related cues, and linked this altered brain activation to relapse risk. Hence, the proposed study will take advantage of the higher spatial resolution and signal-to-noise ratio of a 7 Tesla fMRI scanner to investigate more subtle effects and the involvement of subregions of vlPFC and ACC during alcohol-related inhibition.

Of special interest, particularly when it comes to explaining an imbalance between brain systems related to cue-reactivity and inhibitory control, are concurrent measures of functional brain connectivity. Aberrant resting-state functional connectivity in networks involved in reward prediction, motivation, salience attribution and executive control have been reported in AUD. Also, altered task-related connectivity was observed during cue-reactivity as well as during executive control. However, functional connectivity measures during a task combining both aspects are still missing. Therefore, this study examines the mutual interplay between cue-responsive regions and opposing inhibitory control networks. To this aim, task-related functional connectivity are measured in a specifically tailored experimental design allowing for the assessment of effects related to cue-reactivity, inhibition, as well as their interaction.

Besides, this study assesses whether possible interaction effects of task-related functional connectivity between cue-reactivity and inhibitory control vary with craving, change with prolonged abstinence or predicts drinking outcome.

Taken together, this study will deepen the understanding of the interplay between neuronal networks central to AUD, cue-reactivity and inhibitory control. The (im)balance between these processes is crucial for recently abstinent patients striving to control drinking habits and urges in an environment infused with alcohol-related cues. As such, markers capturing the interaction between these processes are of high conceptual and clinical relevance and might pave the way towards a potential biomarker indicating enhanced relapse risk.

ELIGIBILITY:
Inclusion Criteria:

* Abstained from alcohol for at least 4 weeks prior to fMRI measurement (AUD only)
* Diagnosis of AUD according to ICD-11 (AUD only)
* Written informed consent
* Mother tongue German (or Swiss German)
* Right-handedness
* AUDIT ≤ 7 (HC only)
* AUD-S < 2 (HC only)
* BSCL GSI ≤ 63 (T-value, HC only)
* DUDIT < 7 (HC only)

Exclusion Criteria:

* Other main psychiatric diagnosis than AUD (comorbidity allowed, but AUD has to be considered the main diagnosis, AUD only)
* Neurocognitive problems
* Current medical conditions excluding participation (e.g. acute infectious disease)
* Inability to understand the participant information
* Contraindication to Magnetic Resonance Imaging (e.g. metallic objects, pregnancy, claustrophobia)
* History of alcohol and other substance use disorder (HC only)
* Being staff or student of the project leader and other persons involved in the project

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: AUD patients are detoxified and will be recruited upon entry to specialized residential treatment program at the Clinic Südhang in Kirchlindach in Switzerland.
  HC subjects will be recruited via advertisement in social media and local newspapers in the area of Bern in Switzerland.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-10-13 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
BOLD contrast alcohol vs. neutral inhibition | 3-4 weeks after study inclusion
  The BOLD signal (spatial activation pattern) of alcohol-related stimuli and neutral stimuli during successful inhibition is compared between AUD and HC.
BOLD contrast covariance with craving | 3-4 weeks after study inclusion
  Covariance analysis of the BOLD contrast of successful inhibition between alcohol-related stimuli and neutral stimuli with measures of craving (obsessive compulsive drinking scale, visual analogue scale of craving)

SECONDARY OUTCOMES:
BOLD task-related connectivity | 3-4 weeks after study inclusion
  Psychophysiological interaction (PPI) derived functional connectivity strengths (voxel-to-voxel correlations stratified for cue-type, alcohol vs. neutral), assessing of main effects related to cue-reactivity (alcohol vs. neutral), inhibition (Nogo vs. Go), as well as their interaction and difference between AUD and HC.
BOLD task-related connectivity covariance with craving and drinking outcome | 3 months after GNG-task in fMRI
  Covariance of craving (obsessive compulsive drinking scale, visual analogue scale of craving) and drinking outcome measures (difference in percentage of days abstinent between baseline and 3-month follow-up) with BOLD connectivity of cue-reactivity and inhibitory control.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Grieder, PhD, Principal Investigator — University Hospital for Psychiatry and Psychotherapy Bern
Locations (1):
- University Hospital for Psychiatry and Psychotherapy Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No